CLINICAL TRIAL: NCT03162835
Title: Development and Clinimetric Properties of the Dutch Pediatric Neurophysiology of Pain Questionnaire in Healthy Children
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Roselien Pas, Dra. Roselien Pas, Vrije Universiteit Brussel
Other Study IDs: Eduvalid Study (Part 1)
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Surveys and Questionnaires; Child; Pain; Knowledge; Validation
Keywords: Pain Neuroscience Education
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Educated group: Children within this group will receive Pain Neuroscience Education.
  Interventions: Other: Pain Neuroscience Education
- Non-educated group: Children within this group will not receive Pain Neuroscience Education

INTERVENTIONS:
Other: Pain Neuroscience Education — Children as well as their parents will receive a +/- 1h one-on-one educational session about the neurophysiology of pain, adjusted to the child's comprehension status. Parents will be present in the PNE session too. The PNE program for children contains two sections: (1) The healthy pain system and its function, divided in subsections each consisting of a specific neurophysiological pain concept (i.e. central nervous system anatomy, nociception and nociceptive pathways, up- and down-regulation of the nervous system) and (2) adaptations of the pain system following persistent pain. To ensure interaction between therapist and child, an interactive board game was developed and used throughout the full educational session.
  Groups: Educated group

SUMMARY:
The scientific objective of this research implies developing and examining the clinimetric properties of the Dutch Pediatric Neurophysiology of Pain Questionnaire (PedNPQ) in healthy children.

A total study sample of 60 healthy children (30 from 2nd and 3rd primary school) will be included to measure test-retest reliability of the Pediatric Neurophysiology of Pain Questionnaire (PedNPQ). Children will be asked to fill in the questionnaire twice, with a time interval of 48 hours (assessment T0 and T1).

In order to assess concurrent validity of the PedNPQ, 30 children (15 from 2nd and 3rd primary school) as well as their parent will receive a pediatric Pain Neuroscience Education (PNE) session. It is hypothesized that if the developed PedNPQ is valid, children who received PNE will perform better than children receiving no PNE.

To reduce the participant's workload, all assessments will be done immediately after the school hours or during recreation, in the primary school of the participant.

DETAILED DESCRIPTION:
Pain is a common and daily experience among children that is usually short-term, causing little to moderate discomfort. Yet, a substantial number of children experience chronic pain. Persistent pain periods mainly affect the children's school attendance and participation in recreational activities, possibly leading to academic impairments and social exclusion. Even worse is the children's greater predisposition to develop chronic pain into adulthood. Considering these disadvantages, children suffering from chronic pain should be treated as fast as possible and in the most optimal way. The existing literature on management in children with chronic pain encourages a multidisciplinary approach involving physical therapy and psychological interventions (i.e. cognitive behavioural therapy).

Recently, the application of Pain Neuroscience Education (PNE) as an intervention on its own, as well as in combination with another form of therapy (such as physiotherapy or cognitive- behavioural therapy) is receiving growing interest in the pediatric field of chronic pain. PNE aims to make people understand how their pain is produced and enables them to integrate this understanding into their everyday lives and subsequent treatment components. This innovative education style has shown to be effective in various adult chronic pain populations, by improving the patients' pain coping strategies and health status, and changing their pain beliefs. Although, no study examined the effectiveness of PNE in the context of chronic pediatric pain. The hypothetical efficacy of pediatric PNE is based on previous findings in adult research that a better understanding of the nature of the illness results in improved patient outcomes. When children do not understand the origin of their pain, they might develop irrational beliefs and fears (including catastrophizing) about their pain, sustaining the vicious circle of chronic pain. Indeed, the information and context in which children perceive their pain, has been shown to modulate pain expectations and emotional response to pain. Since research findings showed that even parental beliefs about the aetiology of the child's pain influences the child's pain outcomes, the role of parents as 'pain modulators' might not be underestimated. Therefore, parents should be involved during PNE.

Before and subsequent to providing children and their parents with PNE, it might be interesting to assess their previous knowledge and the change in knowledge about the neurophysiology of pain. To date, this aspect can be evaluated in adults by using the Neurophysiology of Pain Questionnaire (NPQ), a questionnaire developed and published by Moseley et al.. This instrument assesses the patients' reconceptualization of pain, and is validated in English and in Dutch. The questionnaire consists of 19 items and was originally based on examination papers of postgraduate medicine students. Various studies have used the NPQ to evaluated pain-related knowledge in adult chronic pain populations, such as chronic low back pain, chronic fatigue syndrome and chronic whiplash associated disorder. Additionally, previous research suggested the use of the NPQ in a study protocol to evaluate the effectiveness of brief education in the prevention of chronic low-back pain in an at-risk population. Noteworthy, the NPQ is also commonly used in clinical practice as a guideline for clinicians during educational sessions about chronic musculoskeletal pain. Previous research has proven adequate clinimetric properties of the English and Dutch version. One study, using a Rash analysis to evaluate the clinimetric properties of the NPQ in an adult chronic spinal population, found the NPQ to have (1) an acceptable internal consistency to assess individuals, (2) to be effective in targeting the ability of a typical group of chronic pain patients, (3) to be a unidimensional scale and (4) to have good test-retest reliability. Examination of the Dutch version showed fair reliability when retesting occurred within 24 hours, acceptable test-retest reliability and one dimensionality of the questionnaire. To conclude, the NPQ has proven to be a reliable and valid measurement instrument for determining the understanding and knowledge of neurophysiology of pain in adult chronic pain populations and healthcare professionals.

Based on this evidence in adults, it may be valuable to develop and examine the clinimetric properties of a Dutch Pediatric Neurophysiology of Pain Questionnaire (PedNPQ) to determine pain knowledge gaps in children.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children
2. Informed consent

Exclusion Criteria:

1. Previous pain education
2. Chronic pain
3. Insufficient knowledge of the Dutch language
4. Mental retardation
5. Parent with chronic pain

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children will be recruited via announcements in several schools. Children will be eligible for study participation if they meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
Reliability of the Pediatric Neurophysiology of Pain Questionnaire (PedNPQ) | Baseline - 48 hours after baseline
  In order to evaluate test-retest reliability of the test, the two-way mixed infraclass correlation coefficient will be calculated.

SECONDARY OUTCOMES:
Concurrent validity of the Pediatric Neurophysiology of Pain Questionnaire (PedNPQ) | immediately after Pain Neuroscience education (PNE) (48 hours following baseline)
  The validity of the test will be assessed by comparing the test results of the children who received PNE with the children who did not receive PNE.
Responsivity of the Pediatric Neurophysiology of Pain Questionnaire | Baseline, immediately after Pain Neuroscience education (PNE) and 1 week following PNE
  The responsivity of the test will be assessed by comparing the child's baseline responses to the test with their responses after Pain Neuroscience Education.

CONTACTS AND LOCATIONS:
Overall Officials: Roselien Pas, Dra, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Pergolizzi J, Ahlbeck K, Aldington D, Alon E, Coluzzi F, Dahan A, Huygen F, Kocot-Kepska M, Mangas AC, Mavrocordatos P, Morlion B, Muller-Schwefe G, Nicolaou A, Perez Hernandez C, Sichere P, Schafer M, Varrassi G. The development of chronic pain: physiological CHANGE necessitates a multidisciplinary approach to treatment. Curr Med Res Opin. 2013 Sep;29(9):1127-35. doi: 10.1185/03007995.2013.810615. Epub 2013 Jul 3. PMID 23786498
- [Background] Goodman JE, McGrath PJ. The epidemiology of pain in children and adolescents: a review. Pain. 1991 Sep;46(3):247-264. doi: 10.1016/0304-3959(91)90108-A. No abstract available. PMID 1758709
- [Background] Simons LE, Basch MC. State of the art in biobehavioral approaches to the management of chronic pain in childhood. Pain Manag. 2016;6(1):49-61. doi: 10.2217/pmt.15.59. Epub 2015 Dec 17. PMID 26678858
- [Background] Korterink JJ, Diederen K, Benninga MA, Tabbers MM. Epidemiology of pediatric functional abdominal pain disorders: a meta-analysis. PLoS One. 2015 May 20;10(5):e0126982. doi: 10.1371/journal.pone.0126982. eCollection 2015. PMID 25992621
- [Background] Roth-Isigkeit A, Thyen U, Stoven H, Schwarzenberger J, Schmucker P. Pain among children and adolescents: restrictions in daily living and triggering factors. Pediatrics. 2005 Feb;115(2):e152-62. doi: 10.1542/peds.2004-0682. PMID 15687423
- [Background] Vervoort T, Logan DE, Goubert L, De Clercq B, Hublet A. Severity of pediatric pain in relation to school-related functioning and teacher support: an epidemiological study among school-aged children and adolescents. Pain. 2014 Jun;155(6):1118-1127. doi: 10.1016/j.pain.2014.02.021. Epub 2014 Mar 12. PMID 24631587
- [Background] Landry BW, Fischer PR, Driscoll SW, Koch KM, Harbeck-Weber C, Mack KJ, Wilder RT, Bauer BA, Brandenburg JE. Managing Chronic Pain in Children and Adolescents: A Clinical Review. PM R. 2015 Nov;7(11 Suppl):S295-S315. doi: 10.1016/j.pmrj.2015.09.006. PMID 26568508
- [Background] Goddard JM. Chronic pain in children and young people. Curr Opin Support Palliat Care. 2011 Jun;5(2):158-63. doi: 10.1097/SPC.0b013e328345832d. PMID 21415756
- [Background] Robins H, Perron V, Heathcote LC, Simons LE. Pain Neuroscience Education: State of the Art and Application in Pediatrics. Children (Basel). 2016 Dec 21;3(4):43. doi: 10.3390/children3040043. PMID 28009822
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Van Oosterwijck J, Meeus M, Paul L, De Schryver M, Pascal A, Lambrecht L, Nijs J. Pain physiology education improves health status and endogenous pain inhibition in fibromyalgia: a double-blind randomized controlled trial. Clin J Pain. 2013 Oct;29(10):873-82. doi: 10.1097/AJP.0b013e31827c7a7d. PMID 23370076
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Meeus M, Nijs J, Van Oosterwijck J, Van Alsenoy V, Truijen S. Pain physiology education improves pain beliefs in patients with chronic fatigue syndrome compared with pacing and self-management education: a double-blind randomized controlled trial. Arch Phys Med Rehabil. 2010 Aug;91(8):1153-9. doi: 10.1016/j.apmr.2010.04.020. PMID 20684894
- [Background] Jackson T, Pope L, Nagasaka T, Fritch A, Iezzi T, Chen H. The impact of threatening information about pain on coping and pain tolerance. Br J Health Psychol. 2005 Sep;10(Pt 3):441-51. doi: 10.1348/135910705X27587. PMID 16238858
- [Background] Boerner KE, Noel M, Birnie KA, Caes L, Petter M, Chambers CT. Impact of Threat Level, Task Instruction, and Individual Characteristics on Cold Pressor Pain and Fear among Children and Their Parents. Pain Pract. 2016 Jul;16(6):657-68. doi: 10.1111/papr.12306. Epub 2015 May 26. PMID 26011606
- [Background] Palermo TM, Chambers CT. Parent and family factors in pediatric chronic pain and disability: an integrative approach. Pain. 2005 Dec 15;119(1-3):1-4. doi: 10.1016/j.pain.2005.10.027. Epub 2005 Nov 18. No abstract available. PMID 16298492
- [Background] Moseley L. Unraveling the barriers to reconceptualization of the problem in chronic pain: the actual and perceived ability of patients and health professionals to understand the neurophysiology. J Pain. 2003 May;4(4):184-9. doi: 10.1016/s1526-5900(03)00488-7. PMID 14622702
- [Background] Catley MJ, O'Connell NE, Moseley GL. How good is the neurophysiology of pain questionnaire? A Rasch analysis of psychometric properties. J Pain. 2013 Aug;14(8):818-27. doi: 10.1016/j.jpain.2013.02.008. Epub 2013 May 4. PMID 23651882
- [Background] Adillon C, Lozano E, Salvat I. Comparison of pain neurophysiology knowledge among health sciences students: a cross-sectional study. BMC Res Notes. 2015 Oct 22;8:592. doi: 10.1186/s13104-015-1585-y. PMID 26493565
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Moseley GL. Evidence for a direct relationship between cognitive and physical change during an education intervention in people with chronic low back pain. Eur J Pain. 2004 Feb;8(1):39-45. doi: 10.1016/S1090-3801(03)00063-6. PMID 14690673
- [Background] Traeger AC, Moseley GL, Hubscher M, Lee H, Skinner IW, Nicholas MK, Henschke N, Refshauge KM, Blyth FM, Main CJ, Hush JM, Pearce G, McAuley JH. Pain education to prevent chronic low back pain: a study protocol for a randomised controlled trial. BMJ Open. 2014 Jun 2;4(6):e005505. doi: 10.1136/bmjopen-2014-005505. PMID 24889854